CLINICAL TRIAL: NCT07328971
Title: Initial Vancomycin Taper for the Prevention of Recurrent Clostridioides Difficile Infection 2: A Randomized Controlled Trial
Brief Title: Vancomycin Taper to Prevent Recurrent Clostridioides Difficile
Acronym: TAPER-V2
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Emily McDonald, Associate Professor of Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2026-12121
Record Dates: First submitted 2025-11-25; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-11

CONDITIONS: Clostridia Difficile Colitis
Keywords: Clostridoides difficile; Recurrent Clostridioides difficile; C. difficile; Clostridium difficile
MeSH Terms: conditions — Enterocolitis, Pseudomembranous | interventions — Fidaxomicin; Vancomycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fidaxomicin (Active Comparator): Fidaxomicin 200mg PO BID x 10 days
  Interventions: Drug: Fidaxomicin
- Vancomycin T-P (Experimental): Vancomycin 125mg PO QID x2 weeks, then 125mg PO BID x2 weeks, then 125mg PO daily x2 weeks
  Interventions: Drug: Vancomycin capsule

INTERVENTIONS:
Drug: Fidaxomicin — Fidaxomicin 200mg PO BID x 10 days
  Arms: Fidaxomicin
Drug: Vancomycin capsule — Vancomycin 125mg PO QID x2 weeks, then 125mg PO BID x2 weeks, then 125mg PO daily x2 weeks
  Arms: Vancomycin T-P

SUMMARY:
Indirect evidence from network meta-analyses of randomized controlled trials (RCTs) suggest that a pulse and taper (P-T) of vancomycin may be non-inferior to 10-days of fidaxomicin for the prevention of recurrent Clostridioides difficile infections (rCDI). The aim of this trial is:

1) For first episodes and first recurrences of CDI, to test whether a vancomycin P-T is non-inferior to 10-days of fidaxomicin for the prevention of rCDI at 56 days

DETAILED DESCRIPTION:
C. difficile is a gram positive spore-forming anaerobic bacterium that can cause severe diarrhea through colitis. While the incidence of CDI is decreasing in Canada it remains a major cause of both nosocomial and community-acquired diarrhea. The annual incidence of CDI in Canada is 16,000 cases with 1,300 (8.1%) associated deaths. Estimates suggest that CDI is associated with annual economic losses of ~$150 million in Canada and that 23% of these losses are attributable to recurrent cases. Despite appropriate treatment, approximately 20-30% of CDI cases experience a recurrence (rCDI) and recurrent cases are substantially more costly and deadly. Fidaxomicin reduces the absolute recurrence rate of CDI by ~10% relative to 10 days of vancomycin; however, cost and availability prohibit widespread use. At the current price in Canada, fidaxomicin is not cost-effective. Thus, rCDI is associated with significant morbidity, mortality, and economic cost, and prevention is a substantially unmet clinical need.

International CDI guidelines conflict on the recommended treatments for first episodes and first recurrences. The IDSA and ESCMID favor fidaxomicin for both, the ACG recommends fidaxomicin or vancomycin (P-T for first recurrences) for both, whereas the Association of Medical Microbiology and Infectious Disease (AMMI) Canada favors vancomycin for both. These heterogeneous guidelines are mirrored by significant global practice heterogeneity in the use of fidaxomicin or oral vancomycin (10-14 days or as a P-T) for CDI. Since the publication of these guidelines, the TAPER-V trial (NCT04138706) found a 99.0% probability of superiority of a 4-week vancomycin P-T vs. 14 days of vancomycin for first CDI episodes and recurrences for the rCDI outcome at 38 days. Incorporating TAPER-V into a network meta-analysis of RCTs of treatments for first episodes and recurrences revealed that for the prevention of rCDI at day 38, vancomycin P-T was not significantly different from 10 days of fidaxomicin (Adjusted relative risk=0.73, favouring vancomycin P-T, 95% Confidence Interval (95%CI)=0.33, 1.61). However, only indirect evidence was available for this comparison because vancomycin P-T and fidaxomicin have never been compared head-to-head in an RCT.

Although the probability of superiority for vancomycin P-T vs. 14 days of vancomycin in TAPER-V for rCDI was 99.0% at 38 days, this probability fell to 73.8% at 56 days (i.e., the IDSA timeframe for rCDI), and 62.1% at 90 days. All the available RCT evidence for 10 days of fidaxomicin in the prevention of rCDI is within a 40 day timeframe. Thus, it is unknown whether the benefit of fidaxomicin also wanes over time.

By contrast to fidaxomicin, vancomycin P-T has greater worldwide availability and markedly reduced cost. If it is non-inferior or superior to fidaxomicin in terms of preventing rCDI over the long term (e.g., at least 56 days), it will represent a very important addition to international treatment algorithms.

To determine whether vancomycin P-T is an alternative to fidaxomicin, the investigators propose a non-inferiority RCT comparing vancomycin P-T to 10 days of fidaxomicin for the treatment of first episodes and first recurrences of CDI. Indeed, 68.2% of respondents to a recent clinician survey on CDI supported a trial on this comparison. The proposed trial will directly inform clinical practice on the potential of vancomycin P-T as a non-inferior and a lower-cost first-line therapy for CDI. This trial will also be the first to provide data on the longer term rCDI rate (beyond days 38-40) for fidaxomicin.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient or outpatient adults (≥18 years old) treated at the participating institutions.
* First episode or first recurrence of CDI (i.e., second episode within 56 days) defined by a positive C. difficile assay (including PCR toxin gene detection, toxin enzyme immunoassay, and/or cell cytotoxicity neutralization assay37) and the presence of either ≥3 unformed stools in <24 hours with a duration >24 hours, endoscopic/histologic evidence of pseudomembranous colitis, or ileus.
* Because of the prohibitive cost of fidaxomicin, the reimbursement criteria of fidaxomicin by the Régie de l'assurance maladie du Québec will be applied as inclusion criteria until dedicated fidaxomicin funding is available. This includes: either 1) ≥65 years old or immunosuppression, 2) a second episode of C. difficile within 12 weeks of a prior episode of C. difficile, or 3) multiply recurrent CDI (i.e., ≥2 recurrences). When additional funding is obtained, then only inclusion criteria 1 and 2 will be applied.

Exclusion Criteria:

* Planned or current treatment of the present episode of CDI with FMT, intravenous immunoglobulins, or other microbiome therapies (i.e., VOWST or REBYOTA).
* Inability to take medications orally or crushed by tube.
* Prior total colectomy.
* Severe intolerance or allergy to oral vancomycin or fidaxomicin.
* Patient is being admitted to a palliative care ward or is anticipated to die within 3 months of enrollment from another illness.
* Fulminant CDI, defined according to the IDSA definition of CDI with the presence of hypotension, shock, ileus, and/or toxic megacolon. This is because vancomycin is generally preferred at this severity.
* Receipt of more than 72 hours of off-study fidaxomicin or vancomycin CDI therapy for the current episode of CDI.
* Pregnancy or planning to become pregnant during the study period because minimal data on fidaxomicin in pregnancy are available.
* Active breastfeeding because minimal data on fidaxomicin in breastfeeding are available.
* Prior enrollment in this trial.
* Inability to consent without a healthcare proxy.
* Lack of health insurance.
* Anticipated transfer to a site not involved in this trial, or to a palliative care ward.
* Patient declared anticipated inability to participate in study follow-up or lack of means for contact in the outpatient setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
CDI Recurrence | 56 days
  Recurrence will be assessed by clinical record review (chart, laboratory, pharmacy records) and any direct patient interview. CDI recurrence will be defined by 1) three or more unformed stools in a 24-hour period, 2) a positive PCR for toxin gene or and/or detection of toxin by enzyme immunoassay or cell cytotoxicity neutralization assay, and 3) administration of CDI treatment. To avoid missing severe recurrences for cases of ileus, toxic megacolon, or pseudomembranous colitis on colonoscopy the test result and administration of treatment will fulfill criteria for a recurrence in the absence of three or more unformed stools.

SECONDARY OUTCOMES:
All-Cause Mortality | 56 days
  All-cause mortality
All-Cause Mortality | 120 days
  All-cause mortality
Discontinuation of study drug due to adverse events | 56 days
  Discontinuation of the study drug due to any patient-reported adverse event
ER Visit or Hospital (Re)Admission | 56 days
  All-cause ER visits and hospital (re)admission
ER Visit or Hospital (Re)Admission | 120 days
  All-cause ER visits and hospital (re)admission

OTHER OUTCOMES:
Quality of Life: Clostridioides difficile Health-related Quality of Life Questionnaire (Cdiff32) | 56 days
  Patient quality of life will be assessed by the Cdiff32 score value set on enrolment and at day 56; higher scores indicate better health related quality of life.
Quality of life: EuroQol 5 Dimensions 5 Levels (EQ-5D-5L) | 56 days
  patient quality of life will be assessed by the EQ-5D-5L scale Canadian calue set on enrolment and at day 56; higher scores indicate better health status

CONTACTS AND LOCATIONS:
Overall Officials: Emily McDonald, MD MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Todd Lee, MSc MPH, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Louie TJ, Miller MA, Mullane KM, Weiss K, Lentnek A, Golan Y, Gorbach S, Sears P, Shue YK; OPT-80-003 Clinical Study Group. Fidaxomicin versus vancomycin for Clostridium difficile infection. N Engl J Med. 2011 Feb 3;364(5):422-31. doi: 10.1056/NEJMoa0910812. PMID 21288078
- [Background] Johnson S, Lavergne V, Skinner AM, Gonzales-Luna AJ, Garey KW, Kelly CP, Wilcox MH. Clinical Practice Guideline by the Infectious Diseases Society of America (IDSA) and Society for Healthcare Epidemiology of America (SHEA): 2021 Focused Update Guidelines on Management of Clostridioides difficile Infection in Adults. Clin Infect Dis. 2021 Sep 7;73(5):e1029-e1044. doi: 10.1093/cid/ciab549. PMID 34164674
- [Background] McDonald LC, Gerding DN, Johnson S, Bakken JS, Carroll KC, Coffin SE, Dubberke ER, Garey KW, Gould CV, Kelly C, Loo V, Shaklee Sammons J, Sandora TJ, Wilcox MH. Clinical Practice Guidelines for Clostridium difficile Infection in Adults and Children: 2017 Update by the Infectious Diseases Society of America (IDSA) and Society for Healthcare Epidemiology of America (SHEA). Clin Infect Dis. 2018 Mar 19;66(7):e1-e48. doi: 10.1093/cid/cix1085. PMID 29462280